CLINICAL TRIAL: NCT00223184
Title: Study of Prognostic Value by Molecular Analysis in Paediatric Osteosarcomas of the Chromosomal Regions Containing Rb, p16, p53, Cycline D1, APC, erbB2 and C-met Genes
Brief Title: Genetic Characterisation of High-grade Paediatric Osteosarcomas
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Emmanuel LAVOUE, Directeur Adjoint, University Hospital, Strasbourg, France
Other Study IDs: 2472
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Paediatric Osteosarcomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
At present, the only recognised prognostic factor for primary high-grade osteosarcoma is the histological response to preoperative chemotherapy. Our study was designed to identify new diagnostic markers that could eventually have a prognostic value and therapeutic consequences. 80 patients under 20 years of age with primary osteosarcomas were studied while under treatment by the French Society of Paediatric Oncology OS 94 protocol. Paired normal and biopsy samples were collected. In addition, surgical resection specimens, following preoperative chemotherapy, were obtained in many cases. After genomic DNA extraction, an allelotyping analysis targeting microsatellites was planned. The studied DNA regions contained mainly Rb, p53, APC, p16, c-met, TWIST, c-kit, erbB2 and topoisomerases genes. The techniques used in this molecular analysis comprised mainly allelotyping study, quantitative real-time PCR, gene sequencing , immunohistochemistry. The first results showed the prognostic value of 7q31 region containing c-met and 5q21 containing APC (Br J Cancer, 2003, Entz-Werlé et al.), 7p21 containing TWIST (Int J Cancer, 2005, Entz-Werlé et al.) and 4q21 targeting c-kit gene (J Clin Oncol, 2005, Entz-Werlé et al.).

ELIGIBILITY:
Inclusion Criteria:

* Patients under 20 years of age with primary osteosarcomas
* Under treatment by the French Society of Paediatric Oncology OS 94 protocol

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under 20 years of age with primary osteosarcomas
Sampling Method: Non-Probability Sample
Dates: Start 2003-03; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Presence of molecular abnormalities statistically linked to survival or response to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Annie BOILLETOT-BABIN, MD, Principal Investigator — Service de Pédiatrie 3, Hôpital de Hautepierre
Locations (2):
- France (2):
  - Laboratoire de Biologie Moléculaire, Hôpital de Hautepierre, Strasbourg
  - Service de Pédiatrie 3, Hôpital de Hautepierre, Strasbourg